CLINICAL TRIAL: NCT02276014
Title: Effect of SNPs in the Beta-carotene 15, 15'-Monooxygenase (BCMO1) Enzyme on Retinol Formation and Beta-carotene Plasma Responses
Brief Title: Effect of SNPs in the BCMO1 Enzyme
Acronym: BETASNP2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Collaborators: Newcastle University (Other); DSM Nutritional Products, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2011-01-18-BETASNP2; REC 11/NE/0211 (Other: National Research Ethics Service (NRES))
Record Dates: First submitted 2014-10-21; First posted 2014-10-27 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Beta-carotene Bioavailability; Vitamin A Deficiency
Keywords: Beta carotene; Retinol
MeSH Terms: conditions — Vitamin A Deficiency | interventions — beta Carotene

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Supplement A (Other): Beta-carotene 7mg formulation A
  Interventions: Dietary Supplement: Beta-carotene
- Supplement B (Other): Beta-carotene 7mg formulation B
  Interventions: Dietary Supplement: Beta-carotene
- Supplement C (Other): Beta-carotene 7mg formulation C
  Interventions: Dietary Supplement: Beta-carotene

INTERVENTIONS:
Dietary Supplement: Beta-carotene

SUMMARY:
Summary:

Chronic intake of foods low in vitamin A (retinol) and provitamin A forming an unbalanced diet with little variety is common in young individuals in the United Kingdom (UK) population and can lead to subclinical micronutrient deficiency. Provitamin A sources such as β-carotene are cleaved centrally by the β-carotene 15,15'-monooxygenase (BCMO1) into retinal, the precursor of retinol. However, the amount of β-carotene and retinol produced after ingestion of β-carotene is highly variable between healthy individuals, with approximately 40% of the subjects being classified as low responders. Several stable isotope studies have shown a large disparity between the most efficient converters and the most inefficient converters of β-carotene with variations of up to 8-fold. It is possible that differences in β-carotene response may be due to single nucleotide polymorphisms (SNPs) in genes involved in aspects of β-carotene conversion. Previous work has shown that carriers of both, the 379V and 267S+379V BCMO1 variant alleles had a reduced ability to convert β-carotene. More importantly, 44% of the western population have the 379V haplotype. A high percentage of the Western population may therefore not be able to achieve adequate vitamin A intake if dietary β-carotene is a major source of their vitamin A intake. This is of particular relevance to vegetarians, to young individuals aged 19-24 years who have lower intakes of preformed retinol than any other age group, and to pregnant women. The aim of this study is to establish whether the maximum recommended dose for β-carotene of 7mg/day by the British Expert Committee on Vitamins and Minerals (EVM) can overcome the SNP effect in the BCMO1 enzyme.

Hypothesis:

The investigators hypothesize that the current maximum recommended intake of 7 mg of β-carotene per day cannot overcome the low convertor phenotype in BCMO1 to fulfill vitamin A requirements in these people.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individual.
* Female.
* Between 18 and 45 years of age.
* Caucasian.
* BMI between 18 and 30 kg/m2.
* Subject willing and able to give written informed consent.

Exclusion Criteria:

* Smoking.
* Diabetes.
* Gastrointestinal diseases.
* Renal and hepatic diseases.
* Hyperlipidaemia.
* Preformed dietary retinol intake above 60% of reference nutrient intake (RNI) values.
* Recreational drug use.
* Multi-vitamin consumption.
* Pregnancy.
* Menopause.
* Allergy or sensitivity to study products or ingredients.
* Blood donation 3 months prior to screening.
* Participation in other clinical study 4 weeks prior to study start.
* Suspected inability or unwillingness to comply with study procedures.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2012-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of beta-carotene | Pharmacokinetic measures (0,1,4,36,46,57,60 days post-dose)
Area under the plasma concentration versus time curve (AUC) of [13C]retinol | Pharmacokinetic measures (0,1,2,3,4,8,10,22,36,46,57,58,59,60,64,66,78,92,113 days post-dose)

CONTACTS AND LOCATIONS:
Overall Officials: Georg Lietz, PhD, Principal Investigator — Newcastle University
Locations (1):
- Newcastle NIHR Clinical Research Facility, Royal Victoria Infirmary, Newcastle upon Tyne, Tyne & Wear, United Kingdom

REFERENCES:
- [Background] Oxley A, Berry P, Taylor GA, Cowell J, Hall MJ, Hesketh J, Lietz G, Boddy AV. An LC/MS/MS method for stable isotope dilution studies of beta-carotene bioavailability, bioconversion, and vitamin A status in humans. J Lipid Res. 2014 Feb;55(2):319-28. doi: 10.1194/jlr.D040204. Epub 2013 Oct 24. PMID 24158962
- [Background] Lietz G, Oxley A, Leung W, Hesketh J. Single nucleotide polymorphisms upstream from the beta-carotene 15,15'-monoxygenase gene influence provitamin A conversion efficiency in female volunteers. J Nutr. 2012 Jan;142(1):161S-5S. doi: 10.3945/jn.111.140756. Epub 2011 Nov 23. PMID 22113863
- [Background] Grune T, Lietz G, Palou A, Ross AC, Stahl W, Tang G, Thurnham D, Yin SA, Biesalski HK. Beta-carotene is an important vitamin A source for humans. J Nutr. 2010 Dec;140(12):2268S-2285S. doi: 10.3945/jn.109.119024. Epub 2010 Oct 27. PMID 20980645
- [Background] Leung WC, Hessel S, Meplan C, Flint J, Oberhauser V, Tourniaire F, Hesketh JE, von Lintig J, Lietz G. Two common single nucleotide polymorphisms in the gene encoding beta-carotene 15,15'-monoxygenase alter beta-carotene metabolism in female volunteers. FASEB J. 2009 Apr;23(4):1041-53. doi: 10.1096/fj.08-121962. Epub 2008 Dec 22. PMID 19103647
- [Background] Furr HC, Green MH, Haskell M, Mokhtar N, Nestel P, Newton S, Ribaya-Mercado JD, Tang G, Tanumihardjo S, Wasantwisut E. Stable isotope dilution techniques for assessing vitamin A status and bioefficacy of provitamin A carotenoids in humans. Public Health Nutr. 2005 Sep;8(6):596-607. doi: 10.1079/phn2004715. PMID 16236189